CLINICAL TRIAL: NCT01635751
Title: A Randomized, Open-label, 3-way Crossover Clinical Trial to Compare The Pharmacokinetics of A Pregabalin GLARS Tablet 150mg With Immediate Release Formulation and to Assess The Effect of High Fat Diet in Healthy Male Subjects
Brief Title: A Clinical Trial to Compare The Pharmacokinetics of A Pregabalin GLARS Tablet 150mg With Immediate Release Formulation and to Assess The Effect of High Fat Diet in Healthy Male Subjects
Acronym: GLA5PR-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLA5PR-101
Record Dates: First submitted 2012-07-04; First posted 2012-07-10 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Pregabalin; GLARS
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLA5PR GLARS tablet 150mg(fasted) (Experimental)
  Interventions: Drug: Pregabalin
- GLA5PR GLARS tablet 150mg(after high fat meal) (Experimental)
  Interventions: Drug: Pregabalin
- Lyrica Capsule 75mg(fasted) (Active Comparator)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — GLA5PR GLARS tablet 150mg/day(Pregabalin 150mg once a day, fasted)
  Arms: GLA5PR GLARS tablet 150mg(fasted)
Drug: Pregabalin — GLA5PR GLARS tablet 150mg/day(Pregabalin 150mg once a day, after high fat meal)
  Arms: GLA5PR GLARS tablet 150mg(after high fat meal)
Drug: Pregabalin — Lyrica Capsule 150mg/day(Pregabalin 75mg twice a day, fasted)
  Arms: Lyrica Capsule 75mg(fasted)

SUMMARY:
The purpose of this clinical trial is to compare the pharmacokinetic characteristics of GLA5PR GLARS tablet 150mg and Lyrica Capsule 75mg.

GLA5PR GLARS tablet 150mg is a new once-a-day formulation which is made by GL Pharm Tech corporation.

GLARS(Geometrically Long Absorption Regulated System) is new solution to sustained absorption by extending the absorption Site.

To overcome the shortcomings of the currently existing sustained release drug delivery technologies the investigators have recently developed a novel drug delivery system to enable a drug to be dissolved irrespective of the surrounding environment and further absorbed up to colon. The investigators coined this "Geometrically Long Absorption Regulated System(GLARS)".

DETAILED DESCRIPTION:
Basically, this system is a triple-layered tablet, comprised of upper and lower layers that swell and draw a sufficient amount of water, plus a highly water - soluble middle layer that rapidly draw water into the tablet core simultaneously.

The water drawn into the tablet (about 3 to 4 times the weight of the tablet itself) functions as an additional media which enables additional and later drug release out of the dosage form. This serves to overcome the shortage of surrounding media that has been reported to be one of the key reasons for malabsorption of a drug in colon.

As the middle layer induces a rapid water draw into the tablet core, the penetrated water also diffuses to the upper and lower layers, which makes the tablet to rapidly swell and controls drug release.

At virtually the same time, the swollen upper and lower layers form to surround a lateral side of the middle layer, which can, in turn, further control drug release.

This relatively rigid swollen matrix structure makes drug release not affected by surrounding mechanical flux, which can provide relatively consistent in vivo drug release irrespective of degree of gastrointestinal motility.

ELIGIBILITY:
Inclusion Criteria:

* 20~45 years old, Healthy Adult Male Subject
* ≥ 50kg(Body Weight) and Ideal Body Weight ≤ ±20%

Exclusion Criteria:

* ALT or AST > 1.25(Upper Normal Range)
* Total Bilirubin > 1.5 (Upper Normal Range)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cmax | 36hrs
  Pharmacokinetic of Pregabalin
Tmax | 36hrs
  Pharmacokinetic of Pregabalin
AUC0-36h | 36hrs
  Pharmacokinetic of Pregabalin
AUC0-∞ | 36hrs
  Pharmacokinetic of Pregabalin
CL/F | 36hrs
  Pharmacokinetic of Pregabalin
Vd/F | 36hrs
  Pharmacokinetic of Pregabalin
T1/2 | 36hrs
  Pharmacokinetic of Pregabalin

SECONDARY OUTCOMES:
Safety Monitoring | 23 days
  Adverse Event, Vital sign, 12-lead ECG, Laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Dong-seok Yim, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul St.Mary's Hospital, Seochogu, Seoul, South Korea